CLINICAL TRIAL: NCT01417195
Title: A Multicenter, Randomized, Open-label, Parallel-group Study Comparing the Combination of Menopur® and Bravelle® With Menopur® Alone in Subjects Undergoing Assisted Reproductive Technology (ART)
Brief Title: Menopur Mixed Protocol
Acronym: COMBINE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FE999906 CS12
Record Dates: First submitted 2011-07-28; First posted 2011-08-16 (Estimated); Results first posted 2014-04-24 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-05

CONDITIONS: Infertility
Keywords: Assisted Reproductive Technology
MeSH Terms: conditions — Infertility | interventions — Urofollitropin; Menotropins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Menopur and Bravelle combination (Experimental): The initial daily dose consisted of 225 IU of gonadotropins, mixed in the same syringe and administered by subcutaneous (SC) injection for 5 days. The initial daily dose, based on the Investigator's judgment, consisted of either 150 IU of Menopur and 75 IU of Bravelle or 150 IU of Bravelle and 75 IU of Menopur. Dosing adjustments were allowed as of day 6. Dose could vary between 150-450 IU daily and was always to include at least 75 IU of Menopur and 75 IU of Bravelle. Treatment could not continue beyond day 20.
  Interventions: Drug: Bravelle; Drug: Menopur
- Menopur alone (Active Comparator): The initial daily dose consisted of 225 IU of Menopur administered by subcutaneous (SC) injection for 5 days. Dosing adjustments were allowed as of day 6. Dose could vary between 150-450 IU daily and treatment could not continue beyond day 20.
  Interventions: Drug: Menopur

INTERVENTIONS:
Drug: Bravelle
  Other Names: Bravelle®; Urofollitropin; purified form of follicle-stimulating hormone (FSH)
  Arms: Menopur and Bravelle combination
Drug: Menopur
  Other Names: Menopur®; Menotropin; HP-hMG; highly purified menotrophin

SUMMARY:
The objective of this study was to compare the fertilization rate between the combination of Menopur and Bravelle mixed in the same syringe and Menopur alone, both administered subcutaneously (SC), in subjects undergoing Assisted Reproductive Technology (ART). Additionally the study assessed subjects' ability to mix and store the combination of Menopur and Bravelle and to assess safety of the Menopur and Bravelle combination.

ELIGIBILITY:
Main Inclusion Criteria:

* Infertile pre-menopausal female subjects
* Documented history of infertility (eg., unable to conceive for at least 1 year, or 6 months for women ≥36 years of age, or women with bilateral tubal occlusion or absence, or subjects who require donor sperm).
* Subject's male partner with semen analysis that was at least adequate for intracytoplasmic sperm injection (ICSI) within 6 months prior to the subjects beginning down-regulation with gonadotropin-releasing hormone (GnRH)-agonist. Partners with severe male factor requiring invasive or surgical sperm retrieval or donor sperm could have been used.
* Anti-mullerian hormone (AMH) > 1 ng/mL and < 3 ng/mL at screening.
* Eligible for in-vitro fertilisation (IVF) or ICSI treatment.

Main Exclusion Criteria:

* Oocyte donor or embryo recipient; gestational or surrogate carrier
* Previous IVF or assisted reproductive technology (ART) failure due to a poor response to gonadotropins. Poor response was defined as development of ≤ 2 mature follicles or history of 2 previous failed cycle cancellations prior to oocyte retrieval due to poor response.
* Inadequate number of oocytes, defined as fewer than 5 oocytes retrieved in previous ART attempts.
* Subject's male partners with obvious leukospermia (>2 million white blood cells [WBC]/mL) or signs of infection in semen sample within 2 months of the start of subject's pituitary down-regulation. If either of these conditions existed, the male was to be treated with antibiotics and retested prior to subject's pituitary down-regulation.
* Undergoing blastomere biopsy and other experimental ART procedures.
* Body mass index (BMI) of ≤18 and ≥32 kg/m^2

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 122 (Actual)
Dates: Start 2011-07; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (10):
- United States (10):
  - Colorado Center for Reproductive Medicine, Lone Tree, Colorado
  - Women's Medical Research Group, Clearwater, Florida
  - Reproductive Biology Associates, Atlanta, Georgia
  - Fertility Center of Illinois, Chicago, Illinois
  - The Advanced IVF Institute, Naperville, Illinois
  - Shady Grove Fertility, Rockville, Maryland
  - The Center for Assisted Reproduction, Bedford, Texas
  - Houston Fertility Institute, Houston, Texas
  - Center of Reproductive Medicine, Webster, Texas
  - Seattle Reproductive Medicine, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 122 subjects (60 Menopur/Bravelle, 62 Menopur) entered pituitary down-regulation and were randomized in the study.
Period: Overall Study
Arm/Group | Menopur and Bravelle Combination | Menopur Alone
Started | 60 | 62
Completed | 57 | 61
Not Completed | 3 | 1
Not completed — Stimulation failure | 1 | 0
Not completed — No embryos for transfer | 0 | 1
Not completed — No transfer due to risk of OHSS | 1 | 0
Not completed — No transfer due to elevated progesterone | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Menopur Alone: The initial daily dose consisted of 225 IU of Menopur and administered by subcutaneous (SC) injection for 5 days. Dosing adjustments were allowed as of day 6. Dose could vary between 150-450 IU daily and treatment could not continue beyond day 20.
- Total: Total of all reporting groups
Arm/Group | Menopur and Bravelle Combination | Menopur Alone | Total
Number analyzed (Participants) | 60 | 62 | 122
Age, Customized [Number; unit: participants]
  <35 years | 35 | 40 | 75
  35 to 37 years | 13 | 15 | 28
  38 to 40 years | 9 | 6 | 15
  >40 years | 3 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 62 | 122
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White/Caucasian | 42 | 47 | 89
  Black or African American | 9 | 11 | 20
  Asian | 9 | 4 | 13
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic | 6 | 3 | 9
  Non-Hispanic | 54 | 59 | 113
Region of Enrollment [Number; unit: participants]
  United States | 60 | 62 | 122
Body Mass Index [Number; unit: participants]
  18 to <=25 kg/m^2 | 33 | 29 | 62
  >25 to <=30 kg/m^2 | 19 | 23 | 42
  >30 to <=35 kg/m^2 | 8 | 10 | 18
Current Smokers [Number; unit: participants]
  No | 56 | 57 | 113
  Yes | 4 | 5 | 9
Ever Smoked? [Number; unit: participants]
  No | 52 | 56 | 108
  Yes | 8 | 6 | 14
Current Drinkers [Number; unit: participants]
  No | 15 | 11 | 26
  Yes | 45 | 51 | 96

OUTCOME MEASURES:

1. Primary Outcome: Fertilization Rate
Description: The fertilization rate was defined for each participant and calculated as the number of 2 pronuclei (fertilized) (2PN) oocytes divided by the total number of oocytes retrieved multiplied by 100.
Time Frame: approximately day 13 (16-20 hours post insemination by in vitro fertilization (IVF) insemination or intracytoplasmic sperm injection (ICSI))
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: percentage of oocytes retrieved
Arm/Group | Menopur and Bravelle Combination | Menopur Alone
Number analyzed (Participants) | 60 | 62
percentage of oocytes retrieved | 63.14 (21.567) | 59.56 (22.460)
Statistical Analysis 1: Comparison: Menopur and Bravelle Combination vs Menopur Alone; Test type: Non-Inferiority or Equivalence — The pre-defined non-inferiority margin for the lower limit of the 95% CI for the difference in fertilization rate was below -12%; Mean Difference (Final Values) = 3.6, 95% CI 2-sided [-4.3 to 11.5] — Mean difference = Menopur/Bravelle - Menopur. 95% CI is based on Student's t-distribution, assuming equal variances

2. Secondary Outcome: Summary of the Subject Comprehension Questionnaire (SCQ) on Day 1
Description: Subject comprehension questionnaires were completed on Day 1 only by participants assigned to the Menopur and Bravelle treatment arm. On Day 1, the participant read the Mixing Instructions Guide on how to mix and administer the medications at home. The participant was given enough time to read and understand the instructions and ask any questions. The participant then completed the SCQ which consists of 7 questions with YES/NO answers, to self-gauge their understanding of drug administration procedures. Reported data represent the number of participants who answered the question YES. Gonadotropins are referred to as investigational medicinal product (IMP).
Time Frame: Day 1
Population: Intent to treat population for the combination treatment arm only
Measure: Number; unit: participants
Arm/Group | Menopur and Bravelle Combination | Menopur Alone
Number analyzed (Participants) | 60 | 0
participants
  Overall mixing instructions | 60 |
  How to fill the syringe with saline solution | 60 |
  How to mix the first IMP vial with solution | 60 |
  How to mix additional vials of IMP in same syringe | 60 |
  How to inject the IMPs | 60 |
  How to store the IMPs | 60 |
  How to dispose of used vials, syringes, needles | 60 |

3. Secondary Outcome: Summary of the Subject Comprehension Questionnaire (SCQ) on Day 6
Description: Subject comprehension questionnaires were repeated on Day 6 after 5 days of combination therapy by participants assigned to the Menopur and Bravelle treatment arm. The SCQ consists of 7 questions with YES/NO answers to self-gauge participants' understanding of drug administration procedures. Reported data represent the number of participants who answered the question YES. Gonadotropins are referred to as investigational medicinal product (IMP).
Time Frame: Day 6
Population: Intent to treat population for the combination treatment arm only
Measure: Number; unit: participants
Arm/Group | Menopur and Bravelle Combination | Menopur Alone
Number analyzed (Participants) | 60 | 0
participants
  Overall mixing instructions | 60 |
  How to fill the syringe with saline solution | 60 |
  How to mix the first IMP vial with solution | 60 |
  How to mix additional vials of IMP in same syringe | 60 |
  How to inject the IMPs | 60 |
  How to store the IMPs | 60 |
  How to dispose of used vials, syringes, needles | 60 |

4. Secondary Outcome: Summary of Assessor Questionnaire on Day 1
Description: Participants assigned to the Menopur and Bravelle treatment arm read the Mixing Instructions Guide on how to mix and administer the medications at home. Participants were given enough time to read and understand the instructions and ask any questions. After completing the SCQ, participants prepared and self-administered her assigned first daily dose in the presence of the study coordinator or designee assessor. The assessor then completed a 7 question questionnaire with YES or NO answers to document their assessment of participant understanding of drug administration procedures. Reported data represent the number of participants for whom the assessor answered the question YES.
  Gonadotropins are referred to as investigational medicinal product (IMP).
Time Frame: Day 1
Population: Intent to treat population for the combination treatment arm only
Measure: Number; unit: participants
Arm/Group | Menopur and Bravelle Combination | Menopur Alone
Number analyzed (Participants) | 60 | 0
participants
  Acknowledged understanding of mixing instructions | 60 |
  Filled the syringe with saline solution correctly | 60 |
  Mixed the first IMP vial with solution correctly | 60 |
  Mixed additional IMP in same syringe correctly | 60 |
  Injected the IMPs correctly | 60 |
  Acknowledged understanding of how to store IMPs | 60 |
  Disposed used vials, syringes, needles correctly | 60 |

5. Secondary Outcome: Summary of Assessor Questionnaire on Day 6
Description: Participants assigned to the Menopur and Bravelle treatment arm prepared and self-administered her daily dose on Day 6 in the presence of the study coordinator or designee assessor. The assessor then completed a 7 question questionnaire with YES or NO answers to document their assessment of participant understanding of drug administration procedures. Reported data represent the number of participants for whom the assessor answered the question YES.
  Gonadotropins are referred to as investigational medicinal product (IMP).
Time Frame: Day 6
Population: Intent to treat population for the combination treatment arm only
Measure: Number; unit: participants
Arm/Group | Menopur and Bravelle Combination | Menopur Alone
Number analyzed (Participants) | 60 | 0
participants
  Acknowledged understanding of mixing instructions | 60 |
  Filled the syringe with saline solution correctly | 60 |
  Mixed the first IMP vial with solution correctly | 60 |
  Mixed additional IMP in same syringe correctly | 60 |
  Injected the IMPs correctly | 60 |
  Acknowledged understanding of how to store IMPs | 60 |
  Disposed used vials, syringes, needles correctly | 60 |

6. Secondary Outcome: Participants With Treatment Emergent Adverse Events (TEAEs), Including Ovarian Hyperstimulation Syndrome (OHSS)
Description: A treatment-emergent AE was any AE occurring after start of investigational medicinal product (IMP) and within the time of residual drug effect, or a pretreatment AE or pre-existing medical condition that worsened in intensity after start of IMP and within the time of residual drug effect. The time of residual drug effect was the estimated period of time after the last dose of the IMP, where the effect of the product was still considered to be present based on pharmacokinetic, pharmacodynamic, or other IMP characteristics.
Time Frame: Day 1 up to Day 20
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Menopur and Bravelle Combination | Menopur Alone
Number analyzed (Participants) | 60 | 62
participants
  Any TEAEs | 29 | 30
  Drug-related TEAEs | 9 | 13
  Severe TEAEs | 0 | 1
  Serious TEAEs | 0 | 0
  Drug-related Serious TEAEs | 0 | 0
  Any TEAEs resulting in study discontinuation | 0 | 0
  Participants who died | 0 | 0
  Participants with OHSS | 5 | 3
  Cycle cancellation due to OHSS | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 up to Day 20
Arm/Group | Menopur and Bravelle Combination | Menopur Alone
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/62
Other Adverse Events (participants affected / at risk) | 29/60 | 30/62
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Menopur and Bravelle Combination (N=60) | Menopur Alone (N=62)
Abdominal distension (Gastrointestinal disorders) | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 6 | 6
Constipation (Gastrointestinal disorders) | 2 | 3
Nausea (Gastrointestinal disorders) | 2 | 5
Post procedural discomfort (Injury, poisoning and procedural complications) | 2 | 3
Procedural nausea (Injury, poisoning and procedural complications) | 3 | 6
Procedural pain (Injury, poisoning and procedural complications) | 12 | 12
Headache (Nervous system disorders) | 2 | 4
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 5 | 3
Pelvic pain (Reproductive system and breast disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.